CLINICAL TRIAL: NCT06926881
Title: Oscillating Lung Expansion (OLE) Therapy in the Bronchiectasis Patients (BE) Home Care Study Protocol
Brief Title: OLE Therapy With BE Patients in Home Care Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Delve Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BiWaze Clear_001
Record Dates: First submitted 2025-04-08; First posted 2025-04-15 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-04

CONDITIONS: Bronchiectasis; Pulmonary Exacerbation
MeSH Terms: conditions — Bronchiectasis

STUDY DESIGN:
Intervention Model Description: The patient will perform airway clearance therapy with the BiWaze Clear System The BiWaze Clear device includes several components :
  1. BiWaze Clear System. 2. BiWaze Clear Dual Lumen Breathing Circuit. • Dual Lumen bacterial/viral filter. • Dual Lumen breathing tube. • Patient Interface (Anesthesia mask [small, medium or large], Mouthpiece, or trach adapter). 3. Carrying Bag.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- BiWaze Study Device treatment single Arm (Experimental): All patients will be assigned to a single treatment arm utilizing BiWaze Clear System
  Interventions: Device: BiWaze Clear System

INTERVENTIONS:
Device: BiWaze Clear System — The BiWaze Clear device includes several components as follows:
  1. BiWaze Clear System.
  2. BiWaze Clear Dual Lumen Breathing Circuit.
     * Dual Lumen bacterial/viral filter.
     * Dual Lumen breathing tube.
     * Patient Interface (Anesthesia mask [small, medium or large], Mouthpiece, or trach adapter).
  3. Carrying Bag. The patient will perform airway clearance therapy with the BiWaze Clear System

SUMMARY:
The study will examine how the performance of Oscillating Lung Expansion (OLE) therapy affects the respiratory health of patients with Bronchiectasis (BE).

The patient will use the BiWaze Clear system for their airway clearance therapy, instead of their previously prescribed therapy. BiWaze Clear is an FDA-cleared respiratory therapy for assisting patients in loosening and mobilizing secretions as well as treating and preventing atelectasis by providing lung expansion and high-frequency oscillation therapies, combined with aerosol delivery.

The patient will perform airway clearance with BiWaze Clear as prescribed. The system uses a disposable breathing circuit, which is a single patient use, disposable circuit.

The treatment duration is 6 months . The BiWaze Clear System is indicated for the mobilization of secretions, lung expansion therapy, the treatment and prevention of pulmonary atelectasis and has the ability to provide supplemental oxygen when used with an oxygen supply.

DETAILED DESCRIPTION:
The BiWaze Clear System is indicated for the mobilization of secretions, lung expansion therapy, the treatment and prevention of pulmonary atelectasis and has the ability to provide supplemental oxygen when used with an oxygen supply.

The BiWaze Clear System is indicated to deliver therapy to adults and children over the age of 5 years in the home care setting. The primary objective of the study is to evaluate the effectiveness of BiWaze Clear therapy in reducing the frequency of pulmonary exacerbations and improving clinical outcomes.

The study will quantify the frequency of pulmonary exacerbations over a 6-month period during BiWaze Clear therapy and compare this data to the number of exacerbations recorded in the 12 months prior to the initiation of therapy.

A total of 85 adult and pediatric male and female patients (5+ years of age) that are diagnosed with Bronchiectasis(BE) will be enrolled into the study.

The patient will perform airway clearance therapy with the BiWaze Clear System. This system is manufactured by ABM Respiratory Care and assists patients in loosening and mobilizing secretions as well as treating and preventing atelectasis by providing lung expansion and high frequency oscillation therapies. The oscillating lung expansion therapy of the BiWaze Clear System is intended to reduce airway obstructions caused by secretions occupying the lower airways, prevent respiratory tract infections, re-expand the collapsed areas of the lung, thereby enhancing gas exchanges and reducing inflammatory response.

BiWaze Clear provides three respiratory therapies: Positive Expiratory Pressure (PEP), Oscillation (OSC), and Nebulize (NEB).

The study will start with screening patients to confirm eligibility before enrollment Day(-7 to-1). At the screening visit, Informed Consent will be discussed and obtained and signed prior to any study procedures. Potential subjects will be screened by inclusion and exclusion criteria, Medical History and respiratory history will be obtained and documented.

At Visit 1 (Day 1), baseline assessment will be performed, including vital signs, respiratory rate , oxygen saturation, measuring height and weight, recording medical and respiratory history, conduct urine pregnancy test for the female that is able to be pregnant. Bronchiectasis symptoms will be collected , Quality of Life-Bronchiectasis questionnaire will be completed, as well as measuring Forced Expiratory Volume( FEV1) and Forced Vital Capacity (FVC).

Biwaze Clear System Device will be dispensed to the patients. Patients will receive their device training. Remote data-captured devices will be dispensed and provided to the patients along with the respective training.

after the base line visit , there will be another 2 onsite visits where the patients should visit their study sites , Visit 2 ( Day 90) and Visit 3 ( day 180). During these 2 visits, patient's weight will be measured and recorded. V ital signs, respiratory rate, and oxygen saturation will be recorded. Quality of Life-Bronchiectasis questionnaire will be completed, as well as measuring Forced Expiratory Volume( FEV1) and Forced Vital Capacity (FVC). All related AEs and SAEs will be recorded , documented and reported as well as Bronchiectasis symptoms will be collected .

In addition of the screening, baseline visits and onsite visits 2 and 3 , a weekly remote data capture devices will record and report the remote monitoring assessments of study endpoints, including vital signs , respiratory rate, and oxygen saturation, Forced Expiratory Volume( FEV1) and Forced Vital Capacity (FVC) and Bronchiectasis symptoms will be recorded. In addition Quality of Life-Bronchiectasis questionnaire will be completed on a monthly basis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 5 to 85 years old.
2. History of one or more respiratory exacerbations in the past 6 months or two or more respiratory exacerbations in the past 12 months, which required unplanned or unscheduled medical intervention.
3. Ability to perform BiWaze Clear therapy as prescribed.
4. Bronchiectasis diagnosis (including patients with cystic fibrosis with documented bronchiectasis).
5. Signed informed consent (and Child assent if minor subject).

Exclusion Criteria:

1. Diagnosis with rapidly progressing NMD.
2. Post bronchodilator FEV₁ ≥ 65 % predicted
3. Anticipated requirement for hospitalization within the next six months.
4. History of pneumothorax within the past 6 months.
5. Use of OLE therapy within the past 12 months.
6. Inability or unwillingness to perform OLE therapy or study procedures as required.
7. Currently enrolled in a different study.
8. Current smoker or tobacco use within the last 30 days.
9. Pregnancy or Breastfeeding.
10. Any medical conditions deemed by investigators to have a significant impact on the study results, e.g., active cancer, severe cardiovascular, severe progressive pulmonary disease, liver, kidney, or neurological conditions.
11. Inability to comply with the treatment protocol or study procedures.
12. Known allergies to materials used in OLE device.

Ages: 5 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2025-05-20 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate the effectiveness of BiWaze Clear therapy in reducing the frequency of pulmonary exacerbations and improving clinical outcomes. | 6 months
  Quantify the frequency of pulmonary exacerbations over a 6-month period during BiWaze Clear therapy and compare this data to the number of exacerbations recorded in the 12 months prior to the initiation of therapy.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Central Florida Pulmonary Group, P.A., Orlando, Florida
  - Treasure Coast Medical Research Group, LLC, Port Saint Lucie, Florida
  - Metropolitan Clinical Research, Tamarac, Florida
  - University of South Florida -Tampa General Hospital, Tampa, Florida

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: SAP, CSR
Time Frame: Q3-2026